CLINICAL TRIAL: NCT03048344
Title: A Phase I, Two-part Study to Determine the Recommended Dose and Evaluate the Safety and Tolerability of a Novel Oral Arsenic Trioxide Formulation (ORH-2014) in Subjects With Advanced Hematological Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orsenix LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORH2014-001
Record Dates: First submitted 2017-01-31; First posted 2017-02-09 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Advanced Hematological Disorders
Keywords: acute promyelocytic leukemia; APL; arsenic trioxide
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute

STUDY DESIGN:
Intervention Model Description: Part 1 of the study is parallel. Part 2 will be an expansion phase.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental): Subjects will receive oral ORH-2014 at a planned starting dose of 5 mg once daily (QD) in the fasted state. If escalation criteria are met, the administered dose will increase by 5 mg increments to a maximum of 50 mg QD. The starting daily dose is approximately half the typical IV dose (0.15 milligram per kilogram [mg/kg]) extrapolated to a 70-kg person.
  Interventions: Drug: ORH-2014
- Part 2 (Experimental): Subjects will receive a daily oral dose of ORH-2014 at the recommended dose identified in Part 1. ORH-2014 will be administered in the fasted state.
  Interventions: Drug: ORH-2014

INTERVENTIONS:
Drug: ORH-2014 — ORH-2014 capsule 5 mg orally with dose escalations of 5 mg intervals.
  Arms: Part 1
Drug: ORH-2014 — ORH-2014 capsule at recommended dose orally.
  Arms: Part 2

SUMMARY:
Part 1 will be conducted as an open-label, non-randomized, non-placebo-controlled dose escalation study using pre-specified doses. Subjects with the following advanced hematological disorders and no available therapies, and who satisfy all inclusion/exclusion criteria will be enrolled. The purpose is to identify the recommended dose of oral ORH-2014 in subjects with advanced hematological disorders.

Part 2 will be an expansion phase conducted as a single-arm, open-label study to further evaluate the safety and tolerability of ORH-2014 at the maximum tolerated dose (MTD) or recommended dose determined from Part 1 in the fasted state. Subjects with the same disease types as in Part 1 will be enrolled. All subjects will receive oral ORH-2014, in the fasted state, at the recommended dose for an initial period of up to 12 weeks. The purpose is to evaluate the safety and tolerability of oral ORH-2014 in a population of subjects with advanced hematological disorders when administered at the recommended dose.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects ≥18 years of age with one of the following:

  * Relapsed or refractory acute myelocytic leukemia (AML) with nucleophosmin-1 (NPM1) mutations and no available therapies.
  * Relapsed or refractory acute promyelocytic leukemia (APL), with no available therapies. Note: Prior exposure to arsenic trioxide is allowed; however, subjects who have failed arsenic trioxide within the last 12 months are not allowed.
  * Relapsed or refractory myelodysplastic syndrome (MDS), International Prognostic Scoring System intermediate or high-risk, with no available therapies
  * Relapsed or refractory chronic myelomonocytic leukemia (CMML), and other MDS/myeloproliferative neoplasm (MPN) overlap syndromes, with no available therapies
  * Relapsed or refractory mantle cell lymphoma (MCL) with no adequate therapies.
* Negative pregnancy test at the Screening visit for women of childbearing potential and willingness to use adequate birth control
* Not willing to undergo, not a candidate for, or not having a donor for immediate (within 3 months from the Screening date) bone marrow transplantation.

Exclusion Criteria:

* Eastern Cooperative Oncology Group performance status of ≥3;
* Absolute myeloblast count ≥20,000/mm^3;
* Administration of any antineoplastic therapy within 5 half-lives of the antineoplastic therapy before the first dose of ORH-2014, with the exception of hydroxyurea that should be discontinued 1 day prior to the first dose of ORH-2014
* Presence of any remaining toxicities due to previous chemotherapy
* Participation in other clinical trials within at least 2 weeks of the first ORH-2014 dose;
* Clinical evidence of active central nervous system leukemia;
* Active and uncontrolled infection
* Major surgery within 2 weeks prior to trial entry;
* Liver function tests above the following limits at Screening: total bilirubin >1.5 x upper limit of normal (ULN) unless related to Gilbert's syndrome or hemolysis; aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >2.5 x ULN; for subjects with liver involvement, AST and/or ALT >5 x ULN;
* Serum creatinine >1.5 x ULN and/or creatinine clearance or estimated glomerular filtration rate <30 mL/min
* Impaired cardiac function
* Myocardial infarction of unstable angina within 6 months prior to the planned start date of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-12-02 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
To identify the recommended dose | From baseline to Week 4
  The recommended dose is determined by the number of patients who experience a dose limiting toxicity (DLT).
Number of Participants With Adverse Events (AE) as a Measure of Safety and Tolerability of ORH-2014 when administered at the MTD or recommended dose | Up to Week 28
  To evaluate safety and tolerability the aggregate review will include but is not limited to:
  * NCI-CTCAE Grade 3 and 4 AEs, serious adverse events (SAEs), deaths;
  * Laboratory results;
  * Vital signs;
  * ECGs;
  * Individual subject profiles including, but not limited to: medical history, AEs, concomitant medications, laboratory results, and vital signs;
  * Subject disposition and screen failure rates.

SECONDARY OUTCOMES:
To determine the plasma pharmacokinetic (PK) profiles of total arsenic as measured by maximum observed concentration (Cmax) | Baseline up to Week 24
To determine the plasma pharmacokinetic (PK) profiles of total arsenic as measured by time to maximum concentration (Tmax) | Baseline up to Week 24
To determine the plasma pharmacokinetic (PK) profiles of total arsenic as measured by apparent terminal elimination half-life (t1/2) | Baseline up to Week 24
To determine the plasma pharmacokinetic (PK) profiles of total arsenic as measured by area under the concentration-time curve from 0 to 24 hours (AUC0-24) | Baseline up to Week 24
To determine the plasma pharmacokinetic (PK) profiles of total arsenic as measured by area under the concentration-time curve extrapolated to infinity (AUC0-infinity) | Baseline up to Week 24
To determine the plasma pharmacokinetic (PK) profiles of total arsenic as measured by apparent terminal elimination rate constant (λZ) | Baseline up to Week 24
To determine the plasma pharmacokinetic (PK) profiles of total arsenic as measured by apparent total clearance (CL/F) | Baseline up to Week 24
To determine the plasma pharmacokinetic (PK) profiles of total arsenic as measured by apparent total clearance normalized by body weight (CL/F/kg) | Baseline up to Week 24
To determine the plasma pharmacokinetic (PK) profiles of total arsenic as measured by apparent total volume of distribution (Vz/F) | Baseline up to Week 24
To determine the plasma pharmacokinetic (PK) profiles of total arsenic as measured by accumulation ratio (AR) | Baseline up to Week 24
To evaluate the effect of ORH-2014 on QT-interval corrected for heart rate using Fridericia's formula (QTcF) | Baseline up to Week 28
Safety Assessment during the expansion phase of the study on the effect of oral ORH-2014 on safety parameters | Baseline up to Week 28
  During the expansion phase of the study, an aggregate clinical data review (ACDR) will be conducted. This review will collect data from electronic data capture, the ECG central review vendor (ERT), and other sources to include but is not limited to:
  * NCI-CTCAE Grade 3 and 4 AEs, SAEs, deaths;
  * Laboratory results;
  * Vital signs;
  * ECG's;
  * Individual subject profiles including, but not limited to: medical history, AEs, concomitant medications, laboratory results, and vital signs;
  * Subject disposition and screen failure rates.
The number of participants with a complete response (CR) or partial response (PR) according to International Working Group (IWG) response criteria | Up to Week 24
  Bone marrow aspirates and/or biopsies will be obtained at the designated timepoints for evaluation of efficacy. Response criteria will be according to the International Working Group. Responders are participants who obtain complete remission (CR) or partial remission (PR), with or without cytogenetic response, and marrow complete remission.

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, MD, Principal Investigator — MD Anderson
Locations (4):
- United States (4):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Vanderbilt University, Nashville, Tennessee
  - MD Anderson, Houston, Texas

REFERENCES:
- [Derived] Ravandi F, Koumenis I, Johri A, Tallman M, Roboz GJ, Strickland S, Garcia-Manero G, Borthakur G, Naqvi K, Meyer M, Pudipeddi M, Nidarmarthy S, Vaddi K, Kantarjian H. Oral arsenic trioxide ORH-2014 pharmacokinetic and safety profile in patients with advanced hematologic disorders. Haematologica. 2020 Jun;105(6):1567-1574. doi: 10.3324/haematol.2019.229583. Epub 2019 Sep 26. PMID 31558670